CLINICAL TRIAL: NCT04285905
Title: Male Partner-assisted Contact Tracing for HIV and Tuberculosis in Malawi: a Feasibility and Acceptability Study, and Multi-arm Cluster-randomised Trial
Brief Title: Male Partner-assisted Contact Tracing for HIV and Tuberculosis in Malawi
Acronym: mPATCH-TB
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Due to Covid-19, fnding period expired and Phase 2 was not possible.
Sponsor: Liverpool School of Tropical Medicine (Other)
Collaborators: Malawi-Liverpool-Wellcome Trust Clinical Research Programme (Other); London School of Hygiene and Tropical Medicine (Other); University of Liverpool (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 18-020
Record Dates: First submitted 2020-02-24; First posted 2020-02-26 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Tuberculosis
Keywords: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Enhanced standard of care (Active Comparator): * Access to Fast Track TB Clinic
  * Information leaflet for primary male partner
  Interventions: Other: Access to Fast Track TB clinic; Other: Information leaflet for male partner
- Group 2 (Active Comparator): * Access to Fast Track TB Clinic
  * Information leaflet for primary male partner
  * Female participant sputum collection from male partners
  Interventions: Other: Access to Fast Track TB clinic; Other: Information leaflet for male partner; Other: Home sputum collection
- Group 3 (Active Comparator): * Access to Fast Track TB Clinic
  * Information leaflet for primary male partner
  * Female participant sputum collection from male partners
  * Voucher for financial incentive (MKW 5000) that can be collected by the male partner upon attendance at the Fast Track Clinic
  Interventions: Other: Access to Fast Track TB clinic; Other: Information leaflet for male partner; Other: Home sputum collection; Other: Financial incentive
- Group 4 (Active Comparator): * Access to Fast Track TB Clinic
  * Information leaflet for primary male partner
  * Female participant sputum collection from male partners
  * Female partner delivered oral HIV self-testing kits for primary male partner
  Interventions: Other: Access to Fast Track TB clinic; Other: Information leaflet for male partner; Other: Home sputum collection; Other: Home HIV testing
- Group 5 (Active Comparator): * Access to Fast Track TB Clinic
  * Information leaflet for primary male partner
  * Female participant sputum collection from male partners
  * Female partner delivered oral HIV self-testing kits for primary male partner
  * Voucher for financial incentive (MKW 5000) that can be collected by the male partner upon attendance at the Fast Track Clinic
  Interventions: Other: Access to Fast Track TB clinic; Other: Information leaflet for male partner; Other: Home sputum collection; Other: Home HIV testing; Other: Financial incentive

INTERVENTIONS:
Other: Access to Fast Track TB clinic — Male partner can attend clinic with dedicated services for men
Other: Information leaflet for male partner — Female participants will be provided with a letter asking their male partner to attend the clinic for tuberculosis screening
Other: Home sputum collection — Female participants will be provided with sputum cups to take home and collect a sample of sputum from their male partner
  Arms: Group 2; Group 3; Group 4; Group 5
Other: Home HIV testing — Female participants will be provided with an oral HIV self-test kit to be given to their male partner with instructions for use
  Arms: Group 4; Group 5
Other: Financial incentive — Female participants will be provided with a voucher for MKW5000 which can be redeemed when the male partner attends the clinic for TB testing
  Arms: Group 3; Group 5

SUMMARY:
The overall aim of the mPATCH-TB Study is to identify potentially cost-effective, feasible and scalable interventions that could increase rates of completion of screening for tuberculosis and HIV among male partners of women attending primary health care in Blantyre, Malawi.

Eligible women who consent to participate - and who have a primary male partner with cough at home -will be randomly allocated, by day of clinic attendance, into a standard of care group or one of up to four intervention groups. They will be asked to identify their primary male partner and will be offered interventions according to their allocated group.

The primary outcome will compare the proportion of primary male partner that complete TB screening (defined as receipt of result of a sputum Xpert or smear result) within 14 days of recruitment in each intervention group compared to the enhanced standard of care group.

ELIGIBILITY:
Inclusion criteria for female participants

* Female
* Attends study health centre with an acute care episode
* 18 years of age or older on the day of clinic attendance
* Has a primary male partner living within their household
* Reports that primary male partner has symptoms of pulmonary tuberculosis (cough)
* Is resident within urban Blantyre

Inclusion criteria for male partner participants

* Male
* Aged 18 years of age or older on the day of clinic attendance
* Has cough
* Is living with the female participant (defined as sleeping in the same dwelling on most nights during the previous 14 days)

Exclusion criteria for primary male partner participants in trial (applied on the same day the female participant is recruited)

* Currently taking treatment for tuberculosis
* Has taken any treatment for tuberculosis in the 6-months prior to the female participant's clinic attendance
* Is taking isoniazid preventive therapy
* Plans to move out of Blantyre to live elsewhere in the following 2-months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2020-03-28 (Actual); Study Completion 2020-03-28 (Actual)

PRIMARY OUTCOMES:
TB screening | Within 14 days of recruitment of female participant
  The proportion of male partners that complete TB screening

SECONDARY OUTCOMES:
TB case detection | Within 14 days of recruitment of female participant
  The proportion of male partners with either microbiologically-confirmed TB assessment, or taking TB treatment
Acceptability | Within 14 days of recruitment of female participant
  The proportion of primary household male partners who report that they would be "very likely" or "likely" to recommend the interventions they received to their families or friends
Completion of HIV testing | Within 14 days of recruitment of female participant
  The proportion of primary male household partners not receiving ART at baseline who report having been tested for HIV

CONTACTS AND LOCATIONS:
Locations (1):
- Bangwe Health Centre, Blantyre, Southern Region, Malawi

IPD SHARING:
Plan to Share IPD: Yes
To facilitate reproducibility of analysis, an anonymised minimal final dataset and all code required to reproduce analysis will be published in the trial GitHub repository.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: As soon as possible